CLINICAL TRIAL: NCT04360122
Title: Impact of Levamisole and Isoprinosine in Immune-prophylaxis of Egyptian Healthcare Workers Facing COVID-19
Brief Title: Levamisole and Isoprinosine in Immune-prophylaxis of Egyptian Healthcare Workers Facing COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Maged Mohammed Refaat, Professor of Allergy and Clinical Immunology.Faculty of Medicine Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU P20a/ 2020
Record Dates: First submitted 2020-04-15; First posted 2020-04-24 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus Disease (COVID-19)
Keywords: Egypt
MeSH Terms: conditions — COVID-19 | interventions — Levamisole; Inosine Pranobex

STUDY DESIGN:
Intervention Model Description: Phase III, randomized, open labelled, clinical trial on one hundred adult healthy healthcare workers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Levamisole (Active Comparator): Oral Levamisole 150 mg/day for two days per week for two months
  Interventions: Drug: Levamisole
- Isoprinosine (Active Comparator): Oral Isoprinosine 1 g 3 times per day daily for two months
  Interventions: Drug: Isoprinosine
- Levamisole and Isoprinosine (Active Comparator): Oral Levamisole 150 mg/day for two days per week and Oral Isoprinosine 1 g 3 times per day daily for two months
  Interventions: Drug: Levamisole and Isoprinosine
- Non-interventional group (No Intervention): No-intervention

INTERVENTIONS:
Drug: Levamisole — Levamisole (150 mg/day for two days per week for 2 months
  Arms: Levamisole
Drug: Isoprinosine — Isoprinosine (1 g 3 times per day daily) for two months
  Arms: Isoprinosine
Drug: Levamisole and Isoprinosine — Levamisole (150 mg/day for two days per week for 2 months and Isoprinosine (1 g 3 times per day daily) for two months
  Arms: Levamisole and Isoprinosine

SUMMARY:
This randomized open labeled clinical trial will include one hundred healthy healthcare workers who will be randomly assigned into four groups of twenty-five each to receive either levamisole, Isoprinosine, combined levamisole and isoprinosine or no-intervention for two months to detect the impact of Levamisole and Isoprinosine as immune-prophylaxis on the incidence of COVID-19 infection. Participants will be followed-up for three months clinically and laboratory. Blood samples will be collected prior to randomization and during follow up.

DETAILED DESCRIPTION:
One hundred healthy health workers will be randomly assigned to receive either Levamisole, Isoprinosine, Levamisole and Isoprinosine or no-intervention for two months. Written informed consent will be obtained from all participants.

During the study:

1. Participants will be assessed by detailed questionnaire, clinically and laboratory investigations for COVID 19 Detailed questionnaire for: job description, site of isolation hospital, duration of contact, time of exposure, methods of protection Clinically for any symptoms suggestive of COVID19: fever, plus at least one sign or symptom of respiratory disease including cough, shortness of breath, respiratory distress/failure, runny/blocked nose, plus Laboratory: Sampling of the following will be withdrawn from all participants at beginning and end of the study: COVID 19 IgM (for recent infection) or IgG or (old infection)
2. Assessment of the modulatory effect of the drugs will be done by one or more of the following parameters: (at beginning of the study, 2 weeks, 1 month, 2-month, 3 month)

   * Neutrophil function test
   * Natural killer cell count and activity.
   * T cell count and B cell subsets by flowcytometry and activity markers
   * Quantitative immunoglobulines Levels (IgG, IgM, IgA, IgE)
3. Assessment of the drug safety at beginning of the study and every two weeks except for complete blood count every week:

   * Urine analysis
   * Complete blood count with differential to determine total white blood cell count, absolute neutrophilic count (to exclude agranulocytosis) and absolute lymphocytic count (for COVID19).
   * Serum uric acid
   * Renal functions tests
   * Liver function tests

Randomization method:

A block-randomization scheme will be generated by computer software. Computer-generated random numbers will randomize the participants into four intervention groups of 25 each. The patients were randomly assigned to receive either Isoprinosine (1 g 3 times per day daily) or Levamisole (150 mg/day for two days per week), both or no-intervention for two months.

End point of the study:

* Refusal of patient to complete the study.
* Non-compliance on treatment
* Agranulocytosis or thrombocytopenia.
* Hyperuricemia.
* COVID19 infection

ELIGIBILITY:
Inclusion Criteria:

* Adult > 18 years old
* Both Gender (male and female)
* Healthy health care workers employed by one of the hospitals involved in the study
* Negative serology at day 0 for COVID19 infection.
* Evidence of a personally signed and dated informed consent document

Exclusion Criteria:

* Participations in other investigational clinical trials for the treatment or prevention of SARS-COV-2 infection
* Previous or recent COVID 19 infection (previously had a SARS-CoV-2 positive test result or confirmed case of SARS-CoV-2 infection or positive serology at day 0)
* Any medical illness
* Has a congenital immunodeficiency, including specific deficiencies of the interferon-gamma pathway
* Participants receiving steroids, cytotoxic immunosuppressive agents, radiotherapy.
* Participants who have received any other immunotherapy.
* Participants with a history of gout, urolithiasis, nephrolithiasis, renal dysfunction and severe gastric ulcer.
* Participants receiving allopurinol, indomethacin, colchicine or diuretics.
* Participants with hematological problems.
* Known hypersensitivity reactions or Wheat Allergy
* Pregnant and lactating females.
* Refusal to sign the informed consent form
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-20 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Decrease the incidence of COVID-19 infection or its severity | 6 months
  Detect if Levamisole and Isoprinosine can decrease the incidence of COVID-19 infection

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: No